CLINICAL TRIAL: NCT05577260
Title: The Effect of Intraperitoneal Injection of Magnesium Sulphate Versus Dexmedetomidine as an Adjuvant to Bupivacaine on Postoperative Analgesia in Patients Undergoing Abdominal Aortic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, ghada fouad, associate professor of anesthesia, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: -MFM-IRB .R.22.08.1784
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Abdominal Aortic Surgery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D(dexemedetomidine group) (Experimental): Patients receive 20 mL isobaric bupivacaine 0.25% + 1μg/kg Dexmedetomidine completed to 5ml with normal saline.
  Interventions: Drug: Dexmedetomidine; Drug: isobaric bupivacaine
- Group M: (magnesuim sulphate group) (Experimental): Patients received 20ml isobaric bupivacaine 0.25% + 5 ml (500 mg) magnesium sulphate
  Interventions: Drug: magnesuim sulphate; Drug: isobaric bupivacaine

INTERVENTIONS:
Drug: magnesuim sulphate — magnesuim sulphate
  Arms: Group M: (magnesuim sulphate group)
Drug: Dexmedetomidine — Dexmedetomidine
  Arms: Group D(dexemedetomidine group)
Drug: isobaric bupivacaine — 20ml isobaric bupivacaine 0.25%

SUMMARY:
optimal management of postoperative pain is essentiel for better outcome in abdominal aortic surgery.the study aim to compare between analgesic effect of magnesium sulphate versus dexmedetomidine as an adjuvant to bupivacaine when injected intraperitoneal in abdominal aortic surgery.METHODS:50 patients undergoing abdominal aortic surgery are randemelly divided into 2 groups.(group D:patients received 20ml isobaric bupivacaine+1mic/kg dexemedetomidine completed to 5ml normal saline) Group M:patients received 20ml isobaric bupivacaine+5mg magnesuim sulphate .postoperative VAS,MAP will be recorded initially then every 2hours.

DETAILED DESCRIPTION:
AIM OF THE study To compare between analgesic effect of magnesium sulphate versus dexmedetomidine as an adjuvant to bupivacaine when injected intraperitoneal in abdominal aortic surgery methods This study conducted on patients scheduled for abdominal aortic surgery under general anesthesia in Mansoura University Hospitals .The duration of the study is approximately 5 months. The operation will be done after informed written consent from all patients.

Inclusion criteria:

1. Patients scheduled for abdominal aortic surgery under general anesthesia
2. American Society of Anesthesiologists ASA I-III.
3. aged 20-60

Exclusion criteria:

1. Patients with a history of previous abdominal surgery.
2. uncontrolled hypertension or diabetes, major cardiopulmonary disease.
3. psychiatric illness . On the operation day, the patients will be transferred to the operative theater, where a peripheral cannula will be inserted in a suitable forearm vein. All patients received IV midazolam 5 mg to decrease their anxiety. Routine hemodynamic monitoring will be connected, including ECG, pulse oximetry, heart rate, and noninvasive blood pressure.

   We will induce general anesthesia by IV propofol 1-2 mg.kg-1, fentanyl 1 μg.kg-1, in addition to atracurium 0.5 mg.kg-1. Sevoflurane inhalation was used to maintain anesthesia at a minimal alveolar concentration of 2%. Continuous monitoring of hemodynamics was done throughout the procedure. Heart rate and mean arterial pressure (MAP) were recorded at baseline, then every 15 minutes till the operation ended. Hypotension, defined as systolic blood pressure decreased by 20% or more of its baseline value , was managed by crystalloid infusion (5 ml.kg-1) and IV ephedrine (0.1 mg.kg-1). Additionally, bradycardia, defined as heart rate below 50 bpm , was managed by IV atropine (0.2 - 0.5 mg).

   Tested drugs will be prepared in a sterile syringe by the hospital pharmacy and given to the aneasthetist who was blinded to the identity of drugs. After hemostasis was achieved, intraperitoneal instillation of the drugs into the peritoneal cavity by the surgeon.

   After the operation, patients will be transferred to the PACU, then to the internal ward, where close monitoring and assessment will be done. MAP and heart rates were also recorded every 15 minutes for two hours after surgery. They will be instructed to express their pain via the visual analogue score (VAS), with zero for no pain and ten for the maximum pain sensation ever experienced. These readings will be recorded at PACU, then every two hours for the initial 12 hours after surgery, and finally at 16 and 24 hours. If the patient reported a VAS of four or more, IV fentanyl 20-30 μg commenced. The total post-operative opioid consumption was calculated and recorded. Any opioid-related adverse events, including respiratory depression, nausea, and vomiting, were noticed and recorded. The latter two complaints will be managed by IV metoclopramide (10 mg).
4. allergy to study drugs

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for abdominal aortic surgery under general anesthesia
* American Society of Anesthesiologists ASA I-III.

Exclusion Criteria:

* Patients with a history of previous abdominal surgery.
* uncontrolled hypertension or diabetes, major cardiopulmonary disease.
* psychiatric illness .
* allergy to study drugs

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
time for first anelgesic request | 24 hours postoperative
  first postoperative time patients request anelgesia

SECONDARY OUTCOMES:
total anelgesic requirement | 24 hours postoperative
  total dose of anelgesia given to the patients postoperative

CONTACTS AND LOCATIONS:
Overall Officials: GHADA f amer, MD, Principal Investigator — Associate Professor OFanesthesia Mansoura university
Locations (1):
- Mansoura University,Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes